CLINICAL TRIAL: NCT03344770
Title: The Efficacy of Radial Extracorporeal Shockwave Therapy (RESWT) for Functional Improvement of Patients With Knee Osteoarthritis - A Double-blind Randomized Trial
Brief Title: The Efficacy of Radial Extracorporeal Shockwave Therapy on Knee Osteoarthritis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study suspended due to Covid-19 pandemic.
Sponsor: Marta Imamura (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, Principal Investigator, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72067817.8.0000.0068
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rESWT (Experimental): Application of 5,000 pulses of rESWT by a pneumatic generator, with 0.16mJ/mm2 (millijoule per squared millimeter) of energy at a frequency of 20Hz on the most painful spot of the knee. The applications will be given once a week for three weeks.
  Interventions: Device: Active rESWT
- Sham rESWT (Sham Comparator): Application of 5,000 pulses of rESWT by a pneumatic generator, at a frequency of 20Hz on the most painful spot of the knee with 0 mJ/mm2 energy. The applications will also be given once a week for three weeks.
  Interventions: Device: Sham rESWT

INTERVENTIONS:
Device: Active rESWT — 5,000 pulses of rESWT, with 0.16mJ/mm2 of energy at a frequency of 20Hz once a week for three weeks.
  Arms: Active rESWT
Device: Sham rESWT — 5,000 pulses of rESWT, with 0.0 mJ/mm2 of energy at a frequency of 20Hz once a week for three weeks.
  Arms: Sham rESWT

SUMMARY:
This is a double-blind placebo controlled trial whose objective is to understand how much the radial extracorporeal shockwave therapy can improve function of patients with knee osteoarthritis.

For this trial, patients with knee osteoarthritis, after signing the informed consent form and having their demographic and baseline information collected, will be randomly allocated into one of both treatment arms: radial extracorporeal shockwave therapy (rESWT) or sham radial extracorporeal shockwave therapy. Then, they will undertake three sessions of rESWT, for three weeks, i.e. one session per week.

Patients will be assessed prior to the therapy, one week after the end of the therapy and three months after the end of the therapy, and the primary outcome of this study is the functional change measured by the Knee injury and Osteoarthritis Outcome Score (KOOS) validated in Portuguese, three months after the end of the therapy.

Secondary outcomes, will be the change of pain, the change of pressure pain tolerance threshold, change in diffuse noxious inhibitory control (DNIC), and thermographic changes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of knee osteoarthritis;
* Onset knee pain with moderate or severe intensity: Visual Analogue Scale (VAS) > 4;
* Onset knee pain over 3 months prior to the inclusion;

Exclusion Criteria:

* Presence of psychiatric disease;
* Presence of fibromyalgia;
* Presence of systemic inflammatory rheumatic diseases;
* History of neoplasia;
* Presence of clinical diseases in other joints;
* Ongoing use of anticoagulant drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Functional Change | At baseline and three months after the end of the treatment.
  Functional change from baseline, measured by KOOS.

SECONDARY OUTCOMES:
Short Term Functional Changes | At baseline and one week after the end of the treatment.
  Functional change from baseline, measured by KOOS
Knee pain reduction | At baseline, one week and three months after the end of the treatment
  Knee pain changes from baseline, measured by KOOS
Pain pressure threshold tolerance changes | At baseline, one week and three months after the end of the treatment
  Changes in pain pressure threshold tolerance over time, measured by algometer
Diffuse noxious inhibitory control alterations | At baseline, one week and three months after the end of the treatment
  Changes in diffuse noxious inhibitory control over time, measured by algometer
Thermography evaluation | At baseline, one week and three months after the end of the treatment
  Changes thermographic characteristics of lower limbs and knee over time, measured by Infrared Thermography

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Instituto de Medicina Fisica e Reabilitacao HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided